CLINICAL TRIAL: NCT05370352
Title: Effectiveness of Mobile Chat Messaging for Preventing Relapse in Smokers Who Have Recently Quit Smoking: a Randomised Controlled Trial
Brief Title: Mobile Chat Messaging for Smoking Relapse Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government); Tung Wah Group of Hospitals Integrated Centre on Smoking Cessation (Unknown); United Christian Nethersole Community Health Service Smoking Cessation Programme (Unknown)
Responsible Party: Principal Investigator, Tzu Tsun Luk, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19201341
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation
Keywords: relapse prevention; recurrence; mHealth; instant messaging; WhatsApp; chatbot; conversational agent; Chinese
MeSH Terms: conditions — Smoking Cessation; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile chat messaging (Experimental): Standard smoking cessation treatment + Personalised chat messaging
  Interventions: Behavioral: Standard smoking cessation treatment; Behavioral: Personalised chat messaging
- SMS messaging (Active Comparator): Standard smoking cessation treatment + Regular SMS text messaging generic information about the harms of smoking and the benefits of quitting
  Interventions: Behavioral: Standard smoking cessation treatment; Behavioral: SMS text messaging

INTERVENTIONS:
Behavioral: Standard smoking cessation treatment — Standard smoking cessation treatment (behavioural and pharmacotherapy) provided by Tung Wah Group of Hospitals Integrated Centre on Smoking Cessation
Behavioral: Personalised chat messaging — Personalised chat messaging focusing on smoking relapse prevention for 3 months from randomisation. A trained counsellor will interact with a participant individually and provide relapse prevention advice via WhatsApp. The participant can also access a supportive chatbot in WhatsApp, which will provide on-demand smoking relapse prevention support when the counsellor is not available (e.g., during nighttime).
  Arms: Mobile chat messaging
Behavioral: SMS text messaging — SMS text messaging on generic information about the harms of smoking and the benefits of quitting for 3 months from randomisation.
  Arms: SMS messaging

SUMMARY:
Most smokers return to smoking (relapse) after making a quit attempt, but evidence of effective intervention to prevent relapse is scarce. Taking advantage of recent advances in mobile technologies, this study aims to evaluate the effectiveness of a mobile chat messaging-based relapse prevention intervention in promoting successful quitting in people who recently quit smoking (recent abstainers) using a randomised controlled trial design.

DETAILED DESCRIPTION:
Most smokers who made quit attempts and achieved short-term abstinence return to smoking (relapse) over time, even when aided by effective smoking cessation treatment. Since relapse mostly occurred in the first 4 weeks of abstinence, relapse prevention in the early phase of abstinence could potentially boost long-term abstinence. Several behavioural interventions for smoking relapse prevention have been proposed and tested in RCTs. Yet, a 2019 Cochrane review did not find traditional approaches, including self-help materials, telephone counselling and group therapy, effective in increasing long-term abstinence at 6 months or longer.

The widespread use of mobile devices has provided a highly accessible and scalable means for novel behavioural interventions for smoking cessation. A formative qualitative study in current smokers conducted by the investigators showed that mobile chat messaging is a feasible and acceptable platform for delivering smoking cessation support. A subsequent cluster randomised controlled trial on 1148 smokers found that mobile chat messaging combined with brief intervention was effective in increasing biochemically validated abstinence at 6 months. Nonetheless, whether mobile chat messaging could prevent relapse in recent abstainers has remained untested.

The investigators did a pilot trial to confirm the feasibility and acceptability of mobile chat messaging for relapse prevention in recent abstainers. This study aims to evaluate the effectiveness of mobile chat messaging relapse prevention intervention in promoting abstinence in recent abstainers.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 years or above
* Own a smartphone with WhatsApp installed
* Enrolled in a smoking cessation program under Tung Wah Group of Hospitals Integrated Centre on Smoking Cessation
* Smoked daily before the present quit attempt
* Abstained from smoking for 3 to 30 days

Exclusion Criteria:

* Diagnosed with a mental disease or on regular psychotropic drugs
* Participating in other ongoing smoking cessation studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-02-16 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Biochemically validated tobacco abstinence | 6 months after randomisation
  Verified by an exhaled carbon monoxide level of lower than 5 parts per million or a negative salivary cotinine test

SECONDARY OUTCOMES:
Self-reported 6-month prolonged tobacco abstinence | 6 months after randomisation
  Not more than five lapses permitted for 6 months after baseline
Self-reported 7-day point prevalent tobacco abstinence | 3 months after randomisation
  Being completely smoke-free in the past 7 days
Self-reported 7-day point prevalent tobacco abstinence | 6 months after randomisation
  Being completely smoke-free in the past 7 days
Self-reported relapse rate | 3 months after randomisation
  Defined as use of tobacco products for 7 consecutive days or longer
Self-reported relapse rate | 6 months after randomisation
  Defined as use of tobacco products for 7 consecutive days or longer
Biochemically validated tobacco abstinence | 12 months after randomisation
  Verified by an exhaled carbon monoxide level of lower than 5 parts per million or a negative salivary cotinine test
Self-reported 12-month prolonged tobacco abstinence | 12 months after randomisation
  Not more than five lapses permitted for 12 months after baseline
Self-reported 7-day point prevalent tobacco abstinence | 12 months after randomisation
  Being completely smoke-free in the past 7 days
Self-reported relapse rate | 12 months after randomisation
  Defined as use of tobacco products for 7 consecutive days or longer

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Tsun Luk, PhD, RN, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Tung Wah Group of Hospitals Integrated Centre on Smoking Cessation, Hong Kong
  - United Christian Nethersole Community Health Service Smoking Cessation Programme, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Request to obtain IPD can be made to the principal invesitgator on reasonable request

REFERENCES:
- [Background] Luk TT, Wong SW, Lee JJ, Chan SS, Lam TH, Wang MP. Exploring Community Smokers' Perspectives for Developing a Chat-Based Smoking Cessation Intervention Delivered Through Mobile Instant Messaging: Qualitative Study. JMIR Mhealth Uhealth. 2019 Jan 31;7(1):e11954. doi: 10.2196/11954. PMID 30702431
- [Background] Luk TT, Li WHC, Cheung DYT, Wong SW, Kwong ACS, Lai VWY, Chan SS, Lam TH, Wang MP. Chat-based instant messaging support combined with brief smoking cessation interventions for Chinese community smokers in Hong Kong: Rationale and study protocol for a pragmatic, cluster-randomized controlled trial. Contemp Clin Trials. 2019 Feb;77:70-75. doi: 10.1016/j.cct.2018.12.013. Epub 2018 Dec 26. PMID 30593882
- [Background] Wang MP, Luk TT, Wu Y, Li WH, Cheung DY, Kwong AC, Lai V, Chan SS, Lam TH. Chat-based instant messaging support integrated with brief interventions for smoking cessation: a community-based, pragmatic, cluster-randomised controlled trial. Lancet Digit Health. 2019 Aug;1(4):e183-e192. doi: 10.1016/S2589-7500(19)30082-2. Epub 2019 Jul 31. PMID 33323188
- [Background] Luk TT, Cheung YTD, Chan HC, Fok PW, Ho KS, Sze CD, Lam TH, Wang MP. Mobile Chat Messaging for Preventing Smoking Relapse Amid the COVID-19 Pandemic: A Pilot Randomized Controlled Trial. Nicotine Tob Res. 2023 Jan 5;25(2):291-297. doi: 10.1093/ntr/ntac045. PMID 35166327
- [Derived] Luk TT, Su X, Wong V, Chan HC, Wong GN, Lee JKH, Ho SY, Lam TH, Cheung YTD, Wang MP. Mobile Chat Messaging for Smoking Relapse Prevention: A Randomized Clinical Trial. JAMA Intern Med. 2026 Jan 20:e257439. doi: 10.1001/jamainternmed.2025.7439. Online ahead of print. PMID 41557345
- [Derived] Su X, Wong V, Cheung YTD, Chan HC, Wong GN, Lee JKH, Ho SY, Wang MP, Luk TT. Mobile chat messaging for preventing relapse among people who recently quit smoking: Study protocol for a randomized controlled trial. Digit Health. 2024 Oct 21;10:20552076241291709. doi: 10.1177/20552076241291709. eCollection 2024 Jan-Dec. PMID 39439726